CLINICAL TRIAL: NCT05093517
Title: Effect of Novel Glucagon Receptor Antagonist REMD-477 on Glucose and Adipocyte Metabolism in Type 2 Diabetes Mellitus (T2DM)
Brief Title: Effect of Novel Glucagon Receptor Antagonist REMD-477 on Glucose and Adipocyte Metabolism in T2DM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20210463H
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Glucose Tolerance Impaired; Insulin Sensitivity
Keywords: Fasting plasma glucagon; Glucagon receptor antagonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Insulin Resistance | interventions — volagidemab

STUDY DESIGN:
Intervention Model Description: A randomized 2-arm placebo controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded to the study drug or placebo randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glucagon Receptor Agonist (GRA) REMD-477 group (Experimental): Participants are assigned to a 12 week treatment of REMD-477
  Interventions: Drug: REMD-477
- Placebo group (Placebo Comparator): Participants are assigned to a 12 week course of placebo for REMD-477
  Interventions: Drug: Placebo Subcutaneous injection

INTERVENTIONS:
Drug: REMD-477 — A biologic glucagon receptor agonist to which randomized subjects are assigned 2:1
  Arms: Glucagon Receptor Agonist (GRA) REMD-477 group
Drug: Placebo Subcutaneous injection — Placebo for REMD-477 to which subjects will be randomized 1:2.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
With REMD's glucagon receptor antagonist, the study team propose to provide a comprehensive examination of the effect of elevated plasma glucagon concentrations in Type 2 Diabetes Mellitus (T2D) patients on:

(i) glucose tolerance; (ii) insulin sensitivity in liver, muscle, and adipocytes; (iii) beta cell function; (iv) adipocyte inflammation.

DETAILED DESCRIPTION:
Subjects with T2DM inadequately controlled on current medications will participate in a glucose tolerance test, euglycemic insulin clamp combined with 3-3H-glucose and 14-C glycerol infusion, adipose tissue biopsy, before and 12 weeks after treatment with REMD 477 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic subjects, males/females;
2. age = 18-70 years
3. BMI = 25-40 kg/m2;
4. HbA1c = 7.5-10.0%;
5. Type 2 Diabetics who are drug naïve or treated with metformin, sulfonylureas, SGLT-2 inhibitors or any combination thereof.
6. Subjects must be on a stable dose of antidiabetic medications for at least 3 months prior to study.
7. Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
8. Female patients must be non-lactating and must either be at least two years post-menopausal, or be using adequate contraceptive precautions (i.e. oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period

Exclusion Criteria:

1. Subjects with a personal or family history of pancreatic neuroendocrine tumors or multiple endocrine neoplasia, due to the potential increased of pancreatic alpha cell carcinogenicity associated with glucagon receptor antagonists.
2. Subjects with a contraindication to MRI including artificial heart valves or pacemakers
3. Patients with a known sensitivity to humanized antibodies
4. Subjects treated with GLP-1 RAs or insulin are excluded.
5. Subjects treated with a non-antidiabetic medication that may impact insulin sensitivity, such as systemic steroids, or lipase inhibitors (orlistat, Alli or Xenical)
6. Hematocrit < 34 vol%
7. Serum creatinine > 1.8 mg/dl
8. AST (SGOT) > 2 times upper limit of normal
9. ALT (SGPT) > 2 times upper limit of normal
10. Any major organ system disease as identified by medical history, physical exam, and screening blood tests, EKG
11. Subjects who cannot give written, voluntary consent
12. Subjects with a major psychiatric disturbance
13. Only subjects whose body weight has been stable (±3-4 pounds) over the three months prior to study will be included.
14. Patients must not have type 1 diabetes
15. Patients must not have a fasting plasma glucose of greater than 270 mg/dl or HbA1c > 10.0%
16. Patients must not have received a thiazolidinedione, GLP-1 agonist, or insulin for more than one week during the year prior to randomization
17. Patients with a history of clinically significant heart disease (New York Heart Classification greater than class 2; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | Baseline to 13 weeks
  Change in HbA1c measured at baseline and after intervention administration
Fasting Plasma glucose (FPG) | Baseline to 13 weeks
  Change in fasting plasma glucose measured at baseline and after intervention administration
Plasma glucose (PG) | Baseline to 13 weeks
  Change in plasma PG measured at baseline and after intervention administration using an oral glucose tolerance test (OGTT)
Hepatic insulin sensitivity | Baseline to 13 weeks
  Change in hepatic glucose production (HGP)
Whole body glucose disposal | Baseline to 13 weeks
  Change in whole body glucose disposal measured in mg/kg/min
Plasma Free Fatty Acids (FFA) | Baseline to 13 weeks
  Change in plasma free fatty acids
Muscle Insulin sensitivity | Baseline to 13 weeks
  Change in muscle insulin sensitivity measured by insulin-stimulated glucose uptake during low dose high dose insulin clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- Texas Diabetes Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be published in ClinicalTrials.gov as required by law and research findings will be published in a peer reviewed scientific journal.
Supporting Information: Study Protocol
Time Frame: Once the study has completed enrollment and data analysis is complete, data will become available.